CLINICAL TRIAL: NCT02737800
Title: Effect of Prolonged GnRh Agonist Therapy on the Outcome of In-Vitro Fertilization& Embryo Transfer in Endometrioma Patients
Brief Title: Effect of Prolonged GnRh Agonists on Results of Intracytoplasmic Sperm Injection (ICSI ) in Endometrioma Patients
Acronym: GnRh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, lecturer of obgyn., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: obgynivf
Record Dates: First submitted 2016-03-31; First posted 2016-04-14 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Gonadotropin-Releasing Hormone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1A endometrioma more than 5cm (Active Comparator): Endometrioma aspiration GnRh agonist :Decapeptyl 3.75mg intramuscular Standard long stimulation protocol & ICSI
  Interventions: Procedure: endometrioma aspiration; Drug: GnRh agonist ( Decapeptyl ); Procedure: standard long stimulation protocol
- 1B endometrioma more than 5cm control (Sham Comparator): Endometrioma aspiration Standard long stimulation protocol & ICSI
  Interventions: Procedure: endometrioma aspiration; Procedure: standard long stimulation protocol
- 2A endometrioma less than 5cm (Active Comparator): Decapeptyl 3.75mg intramuscular Standard long stimulation protocol & ICSI
  Interventions: Drug: GnRh agonist ( Decapeptyl ); Procedure: standard long stimulation protocol
- 2B endometrioma less than 5cm control (Sham Comparator): Standard long stimulation protocol & ICSI
  Interventions: Procedure: standard long stimulation protocol

INTERVENTIONS:
Procedure: endometrioma aspiration — Transvaginal ultrasound guided aspiration
  Arms: 1A endometrioma more than 5cm; 1B endometrioma more than 5cm control
Drug: GnRh agonist ( Decapeptyl ) — 3 monthly doses of Decapeptyl 7.5mg intramuscular
  Other Names: Decapeptyl
  Arms: 1A endometrioma more than 5cm; 2A endometrioma less than 5cm
Procedure: standard long stimulation protocol — Decapeptyl 3.75mg in the mid luteal phase followed by human menopausal gonadotropins(HMG);fostimon, or merional injections after bleeding, doses are individualization according to each patient, monitored by follicular size &serum estradiol.

SUMMARY:
Investigators compare ICSI results for endometrioma patients with or without cyst aspiration if more than 5cm &with or without GnRh agonists for all endometrioma patients

DETAILED DESCRIPTION:
Group 1 consists of 30 patients of endometrioma more than 5cm subdivided into:

Group 1A;Cyst aspiration followed by standard long protocol in 15 patients Group 1B;Cyst aspiration followed by GnRh suppression for 3 months then standard long protocol in 15 patients

Group 2 consists of 30 patients of endometrioma less than 5cm subdivided into :

Group 2A;no intervention to the cyst. Standard long protocol Group 2B;GnRh suppression for 3 months then standard long protocol

ELIGIBILITY:
Inclusion Criteria:

* endometrioma patients

Exclusion Criteria:

* Follicle stimulating hormone(FSH)10 or more
* hydrosalpinx
* GnRh suppression in the last 12 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with urine pregnancy test positive 2 weeks after embryo transfer | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: suzy abdelaziz, lecturer, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Kasrelaini Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No